CLINICAL TRIAL: NCT05398302
Title: Radiologically Guided Biopsies of Metastatic Castration Resistant Prostate Cancer to Identify Mechanisms of Resistance in Patients Undergoing 177Lu-PSMA Radioligand Therapy
Brief Title: Image-Guided Biopsies to Identify Mechanisms of Resistance in Patients With Metastatic Castration Resistant Prostate Cancer Treated With 177Lu-PSMA Radioligand Therapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-000460; NCI-2021-12416 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-05-23; First posted 2022-05-31 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma; Stage IV Prostate Cancer American Joint Committee on Cancer (AJCC) v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Image-Guided Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (image-guided biopsy) (Experimental): Patients undergo an image-guided biopsy at baseline and 2-4 weeks after cycle 2 of 177Lu-PSMA-617 therapy.
  Interventions: Procedure: Image Guided Biopsy

INTERVENTIONS:
Procedure: Image Guided Biopsy — Undergo image-guided biopsy
  Other Names: Image-Guided Biopsy; Imaging Guided Biopsy

SUMMARY:
This clinical trial studies mechanisms of resistance to 177-lutetium prostate specific membrane antigen (177Lu-PSMA) radioligand therapy using image-guided biopsies in patients with castrate-resistant prostate cancer that had spread to other places in the body (metastatic). Diagnostic procedures, such as image guided biopsies, may help in learning how well 177Lu-PSMA works to kill tumor cells and allow doctors to plan better treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Proportion of metastatic castration resistant prostate cancer (mCRPC) patients with molecular and cellular alterations in tumor, immune and stromal cells after radioligand therapy assessed by histopathology/immunohistochemistry, ribonucleic acid (RNA)-sequencing and proteomic/phospho-proteomic analyses of biopsy samples.

SECONDARY OBJECTIVE:

I. Sequencing to identify frequently mutated genes.

OUTLINE:

Patients undergo an image-guided biopsy at baseline and 2-4 weeks after cycle 2 of 177Lu-PSMA-617 therapy.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer patient
* Histologically confirmed prostate cancer
* Eligible for 177Lu-PSMA-617 under expanded access protocol (IRB# 21-5010) or as part of an approved trial
* Based on positron emission tomography (PET)/computed tomography (CT) images: Evidence of lymph node or soft tissue metastatic disease amenable to image-guided biopsy
* Platelets > 75,000/ul within 14 days prior to biopsy
* Prothrombin time (PT) or International normalized ratio (INR) and a partial thromboplastin time (PTT) < 1.5 times the institutional upper limit normal (ULN) within 14 days prior to biopsy
* Patients on warfarin, aspirin, or other anti-coagulants are eligible provided they are deemed able to tolerate discontinuation of anti-coagulation for one week prior to the biopsy. Conversion to low molecular weight heparin prior to biopsy is permitted per local standard operating procedures, provided there is agreement regarding the procedure between the treating physician, the interventional radiologist and the principal investigator (PI)

Exclusion Criteria:

* Patients with significant congenital or acquired bleeding disorders (e.g. von Wildebrand's disease, acquired bleeding factor inhibitors) are not eligible

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a successful evaluable biopsy with molecular and cellular alterations after radioligand therapy (RLT) | At the end of cycle 2 before the initiation of cycle 3 of RLT (cycle is six weeks)

SECONDARY OUTCOMES:
Proportion of patients with gene mutations that might confer resistance to RLT | At the end of cycle 2 before the initiation of cycle 3 of RLT (cycle is six weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Czernin, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States